CLINICAL TRIAL: NCT00809068
Title: Effects of Tibolone and PPARα-agonist on HDL Metabolism in Postmenopausal Women
Brief Title: High-density Lipoprotein (HDL) Cholesterol in Women Taking Tibolone
Acronym: TibFen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keogh Institute for Medical Research (Other)
Responsible Party: Clinical Professor Bronwyn Stuckey, Keogh Institute for Medical Research
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ID: 2005-001; SCGH Research Grant
Record Dates: First submitted 2008-06-10; First posted 2008-12-16 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: HDL Cholesterol
Keywords: Menopause; menopausal symptoms; tibolone; HDL-C; fenofibrate
MeSH Terms: interventions — Fenofibrate; tibolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): fenofibrate and tibolone
  Interventions: Drug: fenofibrate and tibolone
- 2 (Sham Comparator): tibolone
  Interventions: Drug: tibolone

INTERVENTIONS:
Drug: fenofibrate and tibolone — fenofibrate 160mg daily 8 weeks tibolone 2.5mg daily 23 weeks
  Other Names: Lipidil; Livial
  Arms: 1
Drug: tibolone — tibolone 2.5 mg daily 23 weeks
  Other Names: Livial
  Arms: 2

SUMMARY:
Tibolone (Livial) has been shown in previous studies to lower HDL cholesterol by up to 40%.

This study aims to study the effects of fenofibrate on HDL and subfractions in women taking tibolone.

DETAILED DESCRIPTION:
Tibolone decreases plasma concentrations of HDL cholesterol and HDL-apoA1 and pre-beta HDL, consistent with a pro-atherogenic effect. The mechanism of tibolone on HDL cholesterol has been suggested to result from an acceleration of the catabolism of HDL by stimulation of hepatic lipase with no effect on cellular cholesterol efflux.

PPAR-a agonists, in particular fenofibrate, improve HDL metabolism by increasing the expression and hepatic secretion of HDL apoAI and apoAII.

We hypothesise that fenofibrate will rectify the perturbations on HDL metabolism wrought by tibolone.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* More than 6 months of amenorrhoea
* Raised FSH and low oestradiol level
* If hysterectomised, raised FSH and low oestradiol level

Exclusion Criteria:

* Diabetes
* Renal failure
* Proteinuria
* High alcohol intake
* Regular endurance exercise
* Active weight loss of dieting
* Smokers
* Agents known to influence lipid metabolism
* Major systemic illness
* Intolerance to tibolone and fenofibrate
* Cholelithiasis
* CK and ALT > 2ULN
* Bleeding disorders
* Peptic ulcer disease.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
HDL subpopulation analysis | August 2009

SECONDARY OUTCOMES:
Increase in HDL subpopulations | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn G Stuckey, MBBS FRACP, Principal Investigator — Keogh Institute for Medical Research; Gerald F Watts, MD PhD FRACP, Principal Investigator — School pf Medicine and Pharmacology, Royal Perth Hospital.; Rosalind Hampton, BSc MBBS, Principal Investigator — Keogh Institute for Medical Research; Hugh Barrett, BAgSc PhD, Principal Investigator — School of Medicine and Pharmacology, Royal Perth Hospital
Locations (1):
- Keogh Institute for Medical Research, 'A' Block 3rd Floor, QE II Medical Centre, Nedlands, Perth, Western Australia, Australia